CLINICAL TRIAL: NCT04584255
Title: A Phase II Study of Niraparib With Dostarlimab Therapy as Neoadjuvant Treatment for Patients With BRCA-mutated Breast Cancer
Brief Title: Niraparib + Dostarlimab In BRCA Mutated Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Johns Hopkins University (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-371
Record Dates: First submitted 2020-10-08; First posted 2020-10-12 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; Breast Cancer; HER2-negative Breast Cancer; Germline BRCA1 Gene Mutation; Germline BRCA2 Gene Mutation; Deleterious PALB2 Gene Mutation
Keywords: Invasive Breast Cancer Stage I; Invasive Breast Cancer Stage II; Invasive Breast Cancer Stage III; Breast Cancer; HER2-negative invasive tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — niraparib; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A Triple Negative Breast Cancer (TNBC) (Experimental): Participants will be randomized 1:1 to treatment with the combination (Arm A)
  * Niraparib-Daily beginning with week 1, day 1
  * Dostarlimab-Once every three weeks beginning with week 1, day 1
  Interventions: Drug: Niraparib; Drug: Dostarlimab
- Arm B TNBC (Experimental): Participants will be randomized 1:1 to treatment with the combination (Arm B)
  * 3-week lead-in of niraparib monotherapy followed by treatment with the combination
  * Niraparib Daily beginning with week 1, day 1
  * Dostarlimab Once every three weeks beginning with week 4, day 1
  Interventions: Drug: Niraparib; Drug: Dostarlimab
- Arm C ER+/HER2- (Experimental): exploratory cohort of estrogen receptor (ER) positive HER2-negative participants will be enrolled to Arm C.
  * Niraparib Daily beginning with week 1, day 1
  * Dostarlimab Once every three weeks beginning with week 1, day 1
  Interventions: Drug: Niraparib; Drug: Dostarlimab

INTERVENTIONS:
Drug: Niraparib — Predetermined dosage PO Daily
  Other Names: Zejula
Drug: Dostarlimab — Predetermined Dosage, IV,q3 weeks
  Other Names: TSR042

SUMMARY:
This research study involves pre-operative therapy that is specifically targeted for breast cancer in individuals with BRCA and PALB2 mutations.

The names of the study drugs involved in this study are:

* Niraparib (Zejula)
* Dostarlimab

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including laboratory evaluations, two mandatory research biopsies, imaging assessments, and follow up visits.

Participants will receive treatment for 18 weeks. After 18 weeks, participants will be evaluated to determine if a candidate for surgery or if additional treatment outside of the study.

Participants with triple negative breast cancer will be randomized to one of two treatment arms.

* Arm A: Niraparib with Dostarlimab for 18 weeks
* Arm B: Niraparib alone for 3 weeks, followed by Niraparib with Dostarlimab for 15 weeks

Participants with estrogen receptor positive breast cancer will be placed directly into Arm C. There is no randomization for these participants.

- Arm C: Niraparib with dostarlimab for 18 weeks

It is expected that about 62 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug or drug combination to learn whether the drug combination works in treating a specific disease. "Investigational" means that the study drugs, Niraparib and Dostarlimab, are being studied for use in this setting and the research doctors are trying to learn more about the drug combination-the side effects the combination may cause and if it is effective in treating this type of cancer.

The U.S. Food and Drug Administration (FDA) has not yet approved either of the drugs in this study for your type of cancer. Niraparib has been approved by the FDA for treatment of advanced ovarian cancer in BRCA mutation carriers.

The use of Dostarlimab in this research study is experimental, which means that it is not approved by any regulatory auit is not approved by any regulatory authority, including the FDA, for treatment of breast cancer, or any other disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study. Laboratory assessments for eligibility must be completed within 14 days prior to the date of registration. Diagnostic imaging, such as MRIs and CT scans, must be performed within 28 days of the planned treatment start.
* Participants must have histologically or cytologically confirmed invasive breast cancer Stage I to III with primary tumor size at least 1.0 cm defined by physical exam or imaging (whichever is larger). In the case of a multifocal, multicentric, or bilateral disease, the largest lesion must be ≥ 1.0 cm and designated as the "index" lesion for tumor evaluations. Patients with inflammatory breast carcinoma are not eligible.
* Participants must have documentation of estrogen receptor (ER) and progesterone receptor (PR) testing by IHC according to local institutional guidelines in a CLIA-approved setting. Central confirmation of ER/PR status is not required. All tumors must be HER2 negative.

  * Arms A and B: Target lesion must be ER and PR negative (<10% staining) by local review.
  * Arm C: Target lesion must be ER and/or PR positive (>10% staining) by local review.
* Participants must have documented HER2-negative invasive tumor according to local institutional guidelines in a CLIA-approved setting. Central confirmation of HER2 status is not required. HER2 negative is defined as:

  * 0 or 1+ by IHC, OR
  * Lack of gene amplification with HER2/CEP17 ratio < 2 by ISH, OR
  * Copy number < 6 by ISH
* Participants must have documented germline mutation in BRCA1, BRCA2 or PALB2 that is deleterious or suspected to be deleterious (known or predicted to be detrimental/lead to loss of function). Mutation must be identified through a CLIA-approved laboratory. Final determination of eligibility for any discordant results in pathogenicity will be made by the sponsor-investigator. A formal eligibility exception will not be required in these cases as long as approval by overall study PI is granted and documented.
* Participants with multifocal, multicentric or bilateral disease are eligible if at least one lesion meets criteria for the study. In this circumstance, the investigator must determine which will represent the target lesion to be assessed for response. This should remain consistent throughout the study. The target lesion should be selected on the basis of its size (lesion with the longest diameter) and suitability for accurate repetitive measurements.
* Participants with an eligible target lesion, and another small HER2+ tumor (for example, < 6 mm), may be eligible for enrollment following discussion and agreement with the overall principal investigator. A formal eligibility exception will not be required in these cases as long as approval by the sponsor-investigator is granted and documented.
* Female or male ≥ 18 years of age
* Breast imaging should include imaging of the ipsilateral axilla. For subjects with a clinically positive axilla by physical examination or imaging, axillary tissue acquisition is not required. For patients with a clinically negative axilla by examination and imaging, tissue acquisition is not required. For equivocal imaging findings, tissue acquisition (a needle aspiration, core biopsy) is required. Sentinel Lymph Node (SLN) biopsy before neoadjuvant therapy is not allowed.
* ECOG performance status of 0 or 1
* Adequate organ and bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dl
  * Total serum bilirubin ≤ 1.5 × institutional upper limit of normal (ULN), (≤2.0 in patients with documented Gilbert's Syndrome)
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 × institutional ULN
  * Serum or plasma creatinine ≤ 1.5 × institutional ULN, OR calculated creatinine clearance > 50 mL/min using the Cockcroft-Gault equation
  * International normalized ratio (INR) OR prothrombin time (PT) ≤1.5× ULN. Participants who are receiving anticoagulant therapy are eligible as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) must be ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Premenopausal women must have a negative urine or serum pregnancy test within 7 days of treatment start. Women are considered non-childbearing (by other than medical reasons) if they:

  * are ≥45 years of age and without menses for >1 year
  * have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy with a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * are post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use an adequate barrier method throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Male and female participants of childbearing potential must agree to adhere to adequate contraception as defined in the protocol for the duration of study participation and for 150 days after the last dose of study treatment.
* Female participants must agree to not breastfeed during the study or for 150 days after the last dose of study treatment.
* Participants must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Ability to understand and willingness to sign an informed consent document.
* Ability to swallow and retain oral medication.
* Patients undergoing breast conserving therapy (ie lumpectomy) should not have any contraindications to radiation therapy.
* Participants must be willing to undergo the mandatory research biopsy at baseline and after 3 weeks on study treatment. Participants who undergo an attempted research biopsy procedure for the purpose of this protocol and in whom inadequate tissue is obtained are not required to undergo a repeat biopsy in order to continue on the protocol.

Exclusion Criteria:

* Stage IV breast cancer.
* Concurrent therapy with any other investigational product
* Prior treatment for the current breast cancer, including prior chemotherapy, immune therapy, hormonal therapy, radiation, or investigational therapy for this diagnosis.
* Excisional biopsy of the primary tumor and/or excision of axillary lymph nodes, including SLNB, prior to study treatment.
* Participants with a history of malignancy are ineligible except in the following circumstances:

  * Individuals with a history of invasive breast cancer are not eligible unless they have been disease-free for a minimum of three years.
  * Individuals with a malignancy history other than invasive breast cancer are eligible if they have no active malignancy and are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * Individuals with the following cancer history are eligible: adequately treated nonmelanoma skin cancers, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, stage 1 grade 1 endometrial carcinoma.
  * Other exceptions may exist following agreement with the sponsor-investigator
* Patients with a diagnosis of immunodeficiency, or currently receiving systemic steroid therapy or any other form of immunosuppressive within 7 days prior to the first dose of study treatment. Use of local corticosteroid injections (e.g. intraarticular injections), inhaled, intranasal, ophthalmic, and topical corticosteroids, and subjects requiring corticosteroid pre-medication for hypersensitivity reactions (e.g. CT scan pre-medication) are allowed.
* Patients with autoimmune disease that has required systemic treatment within the past 2 years (i.e. with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Patients with a history of interstitial lung disease or pneumonitis.
* Patients who have received a live vaccine within 2 weeks prior to the start of study treatment.
* Patients who have undergone any major surgery within 3 weeks prior to study entry, patients must have recovered to baseline from any effects of any major surgery.
* Patients with concurrent HIV infection are eligible provided they meet the following criteria:

  * CD4+ T-cell (CD4+) counts ≥ 350 cells/uL
  * No history of AIDS-defining opportunistic infection within 12 months prior to enrollment
  * Any medication used in an antiretroviral therapy (ART) regimen must have no known interaction with the study agents
* Patients with active or chronic Hepatitis B or C are eligible provided they meet the liver function laboratory criteria described in 3.1.10 and cannot be on any medication with a known interaction with the study agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome or psychiatric illness/social situations that would limit compliance with study requirements.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to niraparib, dostarlimab, or their excipients.
* Transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
* Known history of myelodysplastic syndrome (MDS) or or acute myeloid leukemia (AML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2029-07-17 (Estimated)

PRIMARY OUTCOMES:
Tumor-infiltrating lymphocytes (TILs) | baseline to 21 days
  The primary evaluation of change in TILs within each arm will be based on a Wilcoxon signed rank test (absolute difference) using a one-sided alpha = 0.05 for each arm
The number and proportion of participants achieving Pathologic Complete Response (pCR) | 18 weeks
  The number and proportion of participants achieving pCR among all participants who initiate protocol therapy will be summarized with a two-sided 90% exact confidence interval.

SECONDARY OUTCOMES:
pCR rate (ER+/HER2- BC patients) | 18 weeks
  the analysis of pCR will be exploratory and estimation-only, and reported with a two-sided exact 90% confidence interval
Changes in TILs | baseline up to 3 weeks
  Within each arm, the association between changes in TILs and pCR will be evaluated using a two-sample Wilcoxon rank sum test, and the log odds ratio for a fixed change in TILs will be estimated using a simple logistic regression model.
Rate of Residual Cancer Burden (RCB) 0/1 response | 18 Weeks
  Rate of RCB 0/1 response with preoperative combined niraparib and PD-1 blockade in patients with early stage TNBC and ER-positive HER2-negative breast cancer with BRCA-mutations.
  The rate of RCB 0/1 response with preoperative combined niraparib and PD-1 blockade in patients with early stage TNBC (Arm A and B) and ER-positive HER2-negative breast cancer (Arm C) with BRCA-mutations will be estimated and the associated two-sided 90% exact confidence interval will be reported.
Number of Participants With Treatment-Related NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | baseline up to 5 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Erica L. Mayer, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Yale University Cancer Center, New Haven, Connecticut
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dana-farber.org/research/innovations